CLINICAL TRIAL: NCT07300397
Title: Single Patient Investigational Treatment for Cree Leukoencephalopathy (Vanishing White Matter Disease)
Brief Title: Single Patient Investigational Treatment for Cree Leukoencephalopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Genevieve Bernard, MD, MSc, FRCPc, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLE02-ABBV-CLS-7262
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cree Leukoencephalopathy
Keywords: N=1; Cree Leukoencephalopathy; Fosigotifator
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single patient trial (Experimental): Fosigotifator
  Interventions: Drug: Fosigotifator

INTERVENTIONS:
Drug: Fosigotifator — Fosigotifator

SUMMARY:
Cree Leukoencephalopathy (CLE) is a very rare and severe brain disease that mainly affects members of the Cree communities in Northern Quebec. It causes the white matter of the brain-the part that helps nerves communicate-to slowly break down. As the disease progresses, children develop serious neurological problems that worsen over time and, sadly, lead to early death. At the moment, there are no effective treatments for CLE. The disease is caused by a single genetic change in the EIF2B5 gene, the same gene involved in another related condition called Vanishing White Matter (VWM).

A new medication called fosigotifator (FGT, ABBV-CLS-7262) is currently being tested in an international clinical trial for VWM.

The goal of this study is to provide access to this investigational medication (FGT) for a patient with CLE/VWM for whom no other treatment options exist. The study will also look at whether the potential benefits of FGT outweigh the risks, and whether the drug might slow down or stop the brain's white matter from deteriorating. By targeting the underlying cause of the disease, FGT may help reduce neurological symptoms and improve the patient's quality of life.

DETAILED DESCRIPTION:
Cree Leukoencephalopathy (CLE) is a rare and fatal neurodegenerative disorder predominantly affecting the Cree population in Northern Quebec. Characterized by progressive white matter degeneration, this condition leads to severe neurological impairment and decline, leading to premature death. Despite its significant impact on the affected population, there are currently no effective treatments for CLE. CLE is caused by a single founder pathogenic variant in the EIF2B5 gene and is therefore allelic to VWM.

Fosigotifator (FGT, ABBV-CLS-7262) has been developed and its safety and efficacy are currently being studied in a multi-center Phase 1b/2 clinical trial for Vanishing White Matter (VWM) by Calico.

This study aims to provide access to an investigational drug (FGT) for a patient diagnosed with CLE/VWM disease for whom there are no other treatment options available. The study will also evaluate the risk/benefit of FGT in slowing or halting the progression of white matter degeneration in this patient with CLE. By targeting the underlying pathophysiological mechanisms of white matter damage, FGT is expected to alleviate neurological symptoms and improve the quality of life for the patient.

ELIGIBILITY:
Inclusion Criteria:

* • Molecularly confirmed diagnosis of CLE

  * Pre-symptomatic or early symptomatic patient
  * Signed informed consent from the Legal Guardians/caregivers (parents)
  * Must not be eligible for any actively enrolling trial of fosigotifator in CLE/VWM
  * Must be at least 1 month of age at the Baseline visit
  * Must weigh at least 5kg at the Baseline visit

Exclusion Criteria:

* N/A

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2029-01-03 (Estimated); Study Completion 2029-01-03 (Estimated)

PRIMARY OUTCOMES:
Time to death or permanent ventilation | From enrollment to 2 years
  Time to death or permanent ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No